CLINICAL TRIAL: NCT06060756
Title: Assessment of the Occurrence of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) in French Women Suffering from Endometriosis.
Brief Title: Assessment of the Occurrence of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) in Women Suffering from Endometriosis
Acronym: ENDOSAS
Status: Not yet recruiting | Type: Observational
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOSAS
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Endometriosis; Obstructive Sleep Apnea-hypopnea
Keywords: observational; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with confirmed Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) diagnosis: Patients from site's pain unit with confirmed OSAHS diagnosis. OSAHS diagnosis will be made according to standard of care practice in the investigation site, through polysomnography and Epworth Sleepiness Scale (ESS).
  Interventions: Other: questionnaires completion

INTERVENTIONS:
Other: questionnaires completion — Patients will complete the following questionnaires at 3, 6 and 12 months after start of the treatment for Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS):
  * Pain-related questionnaire
  * Endometriosis-specific questionnaire
  * Hospital Anxiety and Depression scale
  * Questionnaire McGill on Quality Of Life
  * Insomnia-related questionnaire

SUMMARY:
This observational study aims at establishing the proportion of patients suffering from endometriosis and for whom an Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) diagnosis is established.

The study participation will be offered to endometriosis patients displaying symptoms that may suggest an underlying OSAHS.

OSAHS diagnosis will be made according to standard of care practice and patients will be followed up to 12 months after initiating the OSAHS treatment to fill in questionnaires assessing the impact of OSAHS treatment on various endometriosis-related symptoms

DETAILED DESCRIPTION:
The overall prevalence of endometriosis varies between 1% and 8% depending on the studies, and endometriosis would affect approximately one in 10 women in France. In 2022, A report was submitted to the President of the French Republic for the development of a national strategy to fight against endometriosis, proposing in particular the development of a national epidemiological database and an "easily identifiable and accessible diagnosis pathway throughout the territory".

The experience at the investigational site has led to note a significant prevalence of obstructive sleep apnea hypopnea syndrome (OSAHS) in the population of patients with endometriosis. There are no published studies on the relationships between OSAHS and endometriosis. However, intermittent hypoxemia and endothelial dysfunction are two important consequences of OSAHS that may be related to endometriosis. Moreover, it is now accepted that OSAHS is correlated with painful bladder syndrome (interstitial cystitis) and the relationship between endometriosis and a decrease in sleep quality as well as chronic fatigue syndrome has also been demonstrated.

Finally, the benefit of Continuous Positive Airway Pressure (CPAP) treatment on endothelial dysfunction has been demonstrated and, empirically, in cooperation with the investigational site's pain unit, a symptomatic improvement in women with endometriosis and OSAHS after initiation of CPAP treatment was observed.

The study aims at exploring the occurrence of OSAHS in patients with endometriosis followed in the site's dedicated pain unit and the impact of OSAHS treatment when it exists, on the symptoms of endometriosis and quality of life.

OSAHS diagnosis will be made according to standard of care practice in the investigation site. Patients with confirmed diagnosis of OSAHS will be treated according to national recommendations for this disease (CPAP or alternative treatments) and will complete questionnaires at 3, 6 and 12 months after start of OSAHS treatment to assess the impact of OSAHS treatment on various endometriosis-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 50 years of age
* Confirmed diagnostic of endometriosis (either through imaging procedure (ultrasound or RMI) or diagnostic coelioscopy)
* Patient suffering from symptoms evocating Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) and justifying a diagnosis process performed within Standard of Care practice
* Patient who has been informed about the study and has signed the informed consent form prior to any study-specific procedures
* Patient willing and able to perform all scheduled procedures in accordance with the study protocol

Exclusion Criteria:

* Post menopausal patient
* Ongoing treatment for OSAHS
* Patient with Chronic Obstructive Pulmonary Disease (COPD) or unstabilized cardiac disorders
* Concomitant participation in another clinical trial
* Pregnant or breastfeeding woman
* Patient under legal protection measure

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with confirmed endometriosis, that are followed for pain at the site's dedicated pain unit, and who display OSAHS symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
the number of patients suffering from endometriosis, followed in the site's dedicated pain unit, and who are diagnosed with Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) | 12 months
  The diagnosis of OSAHS will be performed as per standard of care procedures (medical assessment and polysomnography).Patients with confirmed OSAHS diagnosis will be accounted for the study as positive (Yes) for the primary endpoint.
  Patients who are not diagnosed with OSAHS will be accounted for the study as Negative (No) for the primary endpoint and will discontinue from the study without being followed up to 12 months in the study

SECONDARY OUTCOMES:
Assessment of the impact of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) treatment on endometriosis-associated pain | 3, 6 and 12 months
  Patients with confirmed OSAHS diagnosis will complete Pain-related questionnaire at 3, 6 and 12 months after start of OSAHS treatment
Assessment of the impact of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) treatment on endometriosis-specific symptoms | 3, 6 and 12 months
  Patients with confirmed OSAHS diagnosis will complete Endometriosis-specific questionnaire at 3, 6 and 12 months after start of OSAHS treatment
Assessment of the impact of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) treatment on anxiety and depression | 3, 6 and 12 months
  Patients with confirmed OSAHS diagnosis will complete Hospital Anxiety and Depression scale at 3, 6 and 12 months after start of OSAHS treatment
Assessment of the impact of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) treatment on quality of life | 3, 6 and 12 months
  Patients with confirmed OSAHS diagnosis will complete the Questionnaire McGill on Quality Of Life at 3, 6 and 12 months after start of OSAHS treatment
Exploration of the correlation between answers to the Insomnia-related questionnaire and the sleep disorders objectified by the nocturnal recordings. | 3, 6 and 12 months
  Patients with confirmed OSAHS diagnosis will complete Insomnia Severity Index questionnaire at 3, 6 and 12 months after start of OSAHS treatment
Exploration of the relationship between cardiological symptoms (palpitations, malaise, chest pain) and the existence of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) | 12 months
  Cardiological symptoms occurrence (palpitations, malaise, chest pain) will be assessed from baseline up to the end of study.

IPD SHARING:
Plan to Share IPD: Undecided